CLINICAL TRIAL: NCT00007345
Title: Phase II Trial of Depsipeptide in Patients With Cutaneous T-Cell Lymphoma and Relapsed Peripheral T-Cell Lymphoma
Brief Title: Depsipeptide to Treat Patients With Cutaneous T-Cell Lymphoma and Peripheral T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010049; 01-C-0049; NCT00020436 (obsolete NCT alias)
Record Dates: First submitted 2000-12-16; First posted 2000-12-18 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Cutaneous T Cell Lymphoma; Peripheral T Cell Lymphoma
Keywords: Histone Acetylase; Differentiation; Sezary Syndrome; Mycosis Fungoides; CD 30 Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Sezary Syndrome; Mycosis Fungoides | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Peripheral T-cell Lymphoma (PTCL) (Experimental): Participants received at least one protocol prescribed dose or higher of Romidepsin intravenously at 14mg/m^2 and at 17.5 mg/m^2 on days 1, 8, and 15 of a 28 day cycle.
  Interventions: Drug: Romidepsin
- Cutaneous T-cell Lymphoma (CTCL) (Experimental): Participants received at least one protocol prescribed dose or higher of Romidepsin intravenously at 14mg/m^2 and at 17.5 mg/m^2 on days 1, 8, and 15 of a 28 day cycle.
  Interventions: Drug: Romidepsin

INTERVENTIONS:
Drug: Romidepsin

SUMMARY:
Background:

NSC630176 is a depsipeptide fermentation product from Chromobacterium violaceum with potent cytotoxic activity against human tumor cell lines and in vivo efficacy against both human tumor xenografts and murine tumors (1-3).

NSC 630176, herein referred to as depsipeptide, shows a lack of cross resistance with several commonly used cytotoxic agents such as vincristine, 5-fluorouracil, mitomycin C and cyclophosphamide (2). However, it has been defined as a P-glycoprotein (Pgp) substrate by COMPARE analysis of the National Cancer Institute (NCI) drug screen cytotoxicity profile (4).

Depsipeptide is a member of a novel class of antineoplastic agents, the histone deacetylase inhibitors.

In the phase I trial conducted at the National Cancer Institute (NCI), responses were observed at the maximum tolerated dose (MTD) in patients with cutaneous and peripheral T-cell lymphoma.

Objectives:

In patients with cutaneous T-cell lymphoma, the primary end points to be examined are overall response rate, complete response rate and duration of response.

In patients with relapsed peripheral T-cell lymphoma, the endpoints to be examined are overall response rate and complete response rate.

To evaluate the tolerability of depsipeptide with extended cycles of therapy.

Eligibility:

Patients with cutaneous T-cell lymphoma (mycosis fungoides or Sezary syndrome) or other peripheral T-cell lymphomas are eligible.

Design:

Depsipeptide will be administered at 14 mg/m^2, over 4 hours on days 1, 8 and 15.

This trial will accrue in six cohorts; Arm 1, patients with cutaneous T-cell lymphoma who have had less than or equal to two prior cytotoxic chemotherapy regimens; Arm 2, patients with peripheral T-cell lymphoma who have had less than or equal to two prior cytotoxic chemotherapy regimens; Arm 3, patients with cutaneous and peripheral T-cell lymphoma who have had more than two prior cytotoxic chemotherapy regimens; Arm 4, patients with other mature T-cell lymphomas; Arm 5, a replicate arm of arm 1; Arm 6, patients with peripheral T-cell lymphoma who have had more than two prior cytotoxic chemotherapy regimens; Arm 7, patients with cutaneous T cell lymphoma who have received vorinostat.

Dose may be adjusted based on toxicities.

DETAILED DESCRIPTION:
Background:

NSC630176 is a depsipeptide fermentation product from Chromobacterium violaceum with potent cytotoxic activity against human tumor cell lines and in vivo efficacy against both human tumor xenografts and murine tumors (1-3).

NSC 630176, herein referred to as depsipeptide, shows a lack of cross resistance with several commonly used cytotoxic agents such as vincristine, 5-fluorouracil, mitomycin C and cyclophosphamide (2). However, it has been defined as a P-glycoprotein (Pgp) substrate by COMPARE analysis of the National Cancer Institute (NCI) drug screen cytotoxicity profile (4).

Depsipeptide is a member of a novel class of antineoplastic agents, the histone deacetylase inhibitors.

In the phase I trial conducted at the NCI, responses were observed at the maximum tolerated dose (MTD) in patients with cutaneous and peripheral T-cell lymphoma.

Objectives:

In patients with cutaneous T-cell lymphoma, the primary end points to be examined are overall response rate, complete response rate and duration of response.

In patients with relapsed peripheral T-cell lymphoma, the endpoints to be examined are overall response rate and complete response rate.

To evaluate the tolerability of depsipeptide with extended cycles of therapy.

Eligibility:

Patients with cutaneous T-cell lymphoma (mycosis fungoides or Sezary syndrome) or other peripheral T-cell lymphomas are eligible.

Design:

Depsipeptide will be administered at 14 mg/m^2, over 4 hours on days 1, 8 and 15.

This trial will accrue in six cohorts; Arm 1, patients with cutaneous T-cell lymphoma who have had less than or equal to two prior cytotoxic chemotherapy regimens; Arm 2, patients with peripheral T-cell lymphoma who have had less than or equal to two prior cytotoxic chemotherapy regimens; Arm 3, patients with cutaneous and peripheral T-cell lymphoma who have had more than two prior cytotoxic chemotherapy regimens; Arm 4, patients with other mature T-cell lymphomas; Arm 5, a replicate arm of arm 1; Arm 6, patients with peripheral T-cell lymphoma who have had more than two prior cytotoxic chemotherapy regimens; Arm 7, patients with cutaneous T cell lymphoma who have received vorinostat.

Dose may be adjusted based on toxicities.

ELIGIBILITY:
* INCLUSION CRITERIA:

Based on the Inclusion Criteria outlined below, patients will accrue to one of the cohorts of the trial.

Cohort- chemotherapy regimens allowed. Cohort Status

Cohort 1

Cutaneous T-cell Lymphoma (mycosis fungoides or Sezary syndrome)-2 or fewer. Closed to accrual

Cohort 2

Peripheral T-cell Lymphoma, unspecified, or Anaplastic large cell lymphoma (T and null cell) Primary Cutaneous Type -2 or fewer. Open and accruing

Cohort 3

Cutaneous T-cell Lymphomas or Peripheral T-cell Lymphoma-More than 2. Closed to accrual

Cohort 4

Other Mature T cell Lymphomas-Any number. Open and accruing

Cohort 5

Cutaneous T-cell Lymphoma (mycosis fungoides or Sezary syndrome)-2 or fewer-Cohort 5 is a replicate cohort, identical to #1

Cohort 6

Peripheral T-cell Lymphoma (PTCL), unspecified, or Anaplastic large cell lymphoma (T and null cell) Primary Cutaneous Type-More than 2. Patients with PTCL in cohort 3 migrated to this cohort

Cohort 7

Cutaneous T-cell Lymphoma (mycosis fungoides or Sezary syndrome) Prior vorinostat required-Any number

Patients with cutaneous T-cell lymphoma [CTCL (mycosis fungoides or Sezary syndrome) stage IB to IVB are eligible. Patients with stage IB and IIA should be refractory to, intolerant to, or have reached a six-month or longer response plateau on at least two prior therapies from the following list: psoralen plus ultraviolet A irradiation (PUVA), ultraviolet B (UVB), electron beam therapy (EBT), photophoresis, interferon, systemic cytotoxic chemotherapy, topical nitrogen mustard, or topical carmustine (BCNU). One qualifying prior treatment must have been topical nitrogen mustard, topical carmustine or a phototherapy (UVB, PUVA or EBT). Topical steroids, systemic retinoids or biologicals do not qualify. Patients with stage IB or IIA who are not candidates for topical nitrogen mustard, topical carmustine or phototherapy (UVB, PUVA or EBT) are eligible for enrollment. Patients may not have received more than two systemic cytotoxic chemotherapy regimens. Steroids, retinoids, and biologic agents, will not be considered as systemic cytotoxic chemotherapy. Radiolabeled monoclonal antibody therapy is considered equivalent to a systemic cytotoxic chemotherapy regimen and must be counted toward the two prior systemic cytotoxic regimens. Patients with stage IIB-IVB who have had no more than 2 prior systemic cytotoxic chemotherapeutic regimens are eligible. There is no restriction regarding number of prior topical therapies, skin irradiation, or non-cytotoxic systemic therapies (i.e. PUVA, retinoids or biologic, with the exception of radiolabeled monoclonal antibody therapy) in this patient group. After 24 patients were enrolled in this arm, the arm was closed, and a replicate arm constituted of this same patient population was opened (Cohort 5).

Patients with peripheral T-cell lymphoma (PTCL), unspecified, or anaplastic large cell lymphoma, T and null cell, primary cutaneous type, as defined by the Revised European American Lymphoma (REAL)/World Health Organization (WHO) classification (16-18), who have experienced disease progression after receiving prior standard treatment and who have had no more than 2 prior systemic cytotoxic chemotherapeutic regimens are eligible.

Patients with cutaneous T cell lymphoma (Mycosis fungoides or Sezary Syndrome) or peripheral T cell lymphoma as defined above who have received more than 2 prior systemic therapies and who have experienced disease progression will be included in a third and independent arm. This arm of the protocol was closed to accrual for CTCL with Amendment H.

Patients with mature T cell lymphomas not included above will be enrolled in a fourth arm. These include but are not exclusively limited to: Enteropathy-type T cell lymphoma; Hepatosplenic T-cell lymphoma; Subcutaneous panniculitis-like T cell lymphoma; Angioimmunoblastic T-cell lymphoma; Anaplastic large cell lymphoma. Patients must have experienced disease progression after receiving prior standard treatment. There will be no limit on the number of prior regimens. Primitive T cell neoplasms and T cell leukemias will not be enrolled.

Patients with peripheral T-cell lymphoma, unspecified, or anaplastic large cell lymphoma, T and null cell, primary cutaneous type, as defined by the REAL/WHO classification (16-18), who have experienced disease progression after receiving prior standard treatment and who have had more than 2 prior systemic cytotoxic chemotherapeutic regimens are eligible for enrollment to a sixth arm of the trial.

Patients with cutaneous T cell lymphoma (Mycosis fungoides or Sezary Syndrome) or peripheral T cell lymphoma as defined in #1 who have received any number of prior systemic therapies and who have previously been treated with vorinostat will be included in a third and independent arm. Patients can be enrolled in this arm if they received prior vorinostat and experienced disease progression, subsequent relapse, or had to discontinue to agent due to toxicity.

Disease that is measurable by radiographic imaging, assessing skin lesions, or by quantitating Sezary cell count.

Patients must:

be age greater than or equal to 18 years

have a performance status of Eastern Cooperative Oncology Group (ECOG) 0-2

have no serious or intercurrent illness and have a life expectancy of greater than 12 weeks

give written informed consent

female patients of childbearing potential must have a negative pregnancy test within 4 weeks and must use effective contraception

sexually active males must use effective contraception

Laboratory values (performed less than or equal to 14 days prior to registration):

absolute neutrophil count greater than or equal to 1000/microliter, platelets greater than or equal to l00,000/microliter, bilirubin (total and direct) less than or equal to 1.5x upper limit of normal, and aspartate aminotransferase (AST) less than or equal to 3x upper limit of normal, unless impairment is due to organ involvement by lymphoma, creatinine less than or equal to 1.5x upper limit of normal, or documented creatinine clearance of greater than or equal to 60mL/min

Cardiac studies (performed within 4 weeks of registration):

Ejection fraction of greater than 50% by Echocardiogram or Cardiac magnetic resonance imaging (MRI), or greater than or equal to 45% by multi-gated acquisition scan (MUGA) Scan.

A stable dose (greater than 1 month) of corticosteroids administered for symptom management will not preclude enrollment. Tapering will be initiated following administration of depsipeptide.

EXCLUSION CRITERIA:

Patients with unconfirmed diagnosis, or with B-cell lymphomas will be excluded.

Prior or concurrent malignancies that have not been curatively treated.

Known central nervous system (CNS) lymphoma.

Chemotherapy within 4 weeks, 6 weeks for nitrosoureas or mitomycin C.

Biologics, Immunotherapy within 2 weeks.

Human Immunodeficiency virus (HIV) seropositivity.

Pregnant or breast-feeding patients.

Major surgery within 21 days.

Uncontrolled infection or uncontrolled medical illness.

Patients having received prior histone deacetylase (HDAC) inhibitor therapy for T cell lymphoma will be excluded except for patients eligible to enroll in cohort 7.

Patients with the following cardiac risk factors will be excluded from the study:

Patients with known cardiac abnormalities such as:

Congenital long QT syndrome

Corrected QT interval (QTc) interval greater than 480 milliseconds

Patients who have had a myocardial infarction within 12 months of study entry.

Patients who have active coronary artery disease as, e.g. angina as defined by Canadian Class II-IV

Patients with an electrocardiography (ECG) recorded at screening showing evidence of cardiac ischemia (ST depression of greater than or equal to 2 mm).

Any patient in whom coronary artery disease is suspected should be referred for a cardiology consultation and if active myocardial ischemia is demonstrated the patient should be excluded. If a noninvasive imaging study is equivocal, it may be necessary to proceed to coronary angiography.

Patients with congestive heart failure that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction less than 45% by MUGA scan or less than 50% by echocardiogram and/or MRI.

Patients with a history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD). Patients with a history of arrhythmia should have Holter monitoring and evaluation by cardiology.

Patients with dilated, hypertrophic, or restrictive cardiomyopathy from prior treatment or other causes (in doubt, see ejection fraction criteria above). Patients with left ventricular hypertrophy should be discussed with the Principal Investigator or Study Chairman.

Patients with uncontrolled hypertension, i.e., systolic blood pressure (SBP) greater than or equal to 160 mm Hg or diastolic blood pressure (DBP) greater than or equal to 95 mm Hg.

Patients with cardiac arrhythmia requiring anti-arrhythmic medication other than beta blocker or calcium channel blocker. Patients in whom digitalis cannot be discontinued are excluded from study.

Patients with Mobitz II second degree heart block who do not have a pacemaker. Patients with first degree or Mobitz I second degree heart block, bradyarrhythmias or sick sinus syndrome require Holter monitoring and evaluation by cardiology.

Patients with other cardiac disease may be excluded at the discretion of the principal investigator (PI) following consultation with cardiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2001-03-08 (Actual); Primary Completion 2015-01-26 (Actual); Study Completion 2015-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (13):
- United States (10):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - City of Hope National Cancer Center, Duarte, California
  - Mercy General Hospital, Sacramento, California
  - Georgetown University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - North Shore University Hospital, Manhasset, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - West Virginia University, Morgantown, West Virginia
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Peter MacCallum Cancer Centre, Melbourne
  - Sir Charles Gairdner Hospital, Perth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piekarz RL, Frye AR, Wright JJ, Steinberg SM, Liewehr DJ, Rosing DR, Sachdev V, Fojo T, Bates SE. Cardiac studies in patients treated with depsipeptide, FK228, in a phase II trial for T-cell lymphoma. Clin Cancer Res. 2006 Jun 15;12(12):3762-73. doi: 10.1158/1078-0432.CCR-05-2095. PMID 16778104
- [Background] Woo S, Gardner ER, Chen X, Ockers SB, Baum CE, Sissung TM, Price DK, Frye R, Piekarz RL, Bates SE, Figg WD. Population pharmacokinetics of romidepsin in patients with cutaneous T-cell lymphoma and relapsed peripheral T-cell lymphoma. Clin Cancer Res. 2009 Feb 15;15(4):1496-503. doi: 10.1158/1078-0432.CCR-08-1215. PMID 19228751
- [Background] Ritchie D, Piekarz RL, Blombery P, Karai LJ, Pittaluga S, Jaffe ES, Raffeld M, Janik JE, Prince HM, Bates SE. Reactivation of DNA viruses in association with histone deacetylase inhibitor therapy: a case series report. Haematologica. 2009 Nov;94(11):1618-22. doi: 10.3324/haematol.2009.008607. Epub 2009 Jul 16. PMID 19608677
- [Background] Bates SE, Zhan Z, Steadman K, Obrzut T, Luchenko V, Frye R, Robey RW, Turner M, Gardner ER, Figg WD, Steinberg SM, Ling A, Fojo T, To KW, Piekarz RL. Laboratory correlates for a phase II trial of romidepsin in cutaneous and peripheral T-cell lymphoma. Br J Haematol. 2010 Jan;148(2):256-67. doi: 10.1111/j.1365-2141.2009.07954.x. Epub 2009 Oct 28. PMID 19874311
- [Background] Akilov OE, Grant C, Frye R, Bates S, Piekarz R, Geskin LJ. Low-dose electron beam radiation and romidepsin therapy for symptomatic cutaneous T-cell lymphoma lesions. Br J Dermatol. 2012 Jul;167(1):194-7. doi: 10.1111/j.1365-2133.2012.10905.x. PMID 22372971
- [Background] Noonan AM, Eisch RA, Liewehr DJ, Sissung TM, Venzon DJ, Flagg TP, Haigney MC, Steinberg SM, Figg WD, Piekarz RL, Bates SE. Electrocardiographic studies of romidepsin demonstrate its safety and identify a potential role for K(ATP) channel. Clin Cancer Res. 2013 Jun 1;19(11):3095-104. doi: 10.1158/1078-0432.CCR-13-0109. Epub 2013 Apr 15. PMID 23589175
- [Result] Bates SE, Eisch R, Ling A, Rosing D, Turner M, Pittaluga S, Prince HM, Kirschbaum MH, Allen SL, Zain J, Geskin LJ, Joske D, Popplewell L, Cowen EW, Jaffe ES, Nichols J, Kennedy S, Steinberg SM, Liewehr DJ, Showe LC, Steakley C, Wright J, Fojo T, Litman T, Piekarz RL. Romidepsin in peripheral and cutaneous T-cell lymphoma: mechanistic implications from clinical and correlative data. Br J Haematol. 2015 Jul;170(1):96-109. doi: 10.1111/bjh.13400. Epub 2015 Apr 19. PMID 25891346
- [Result] Piekarz RL, Frye R, Turner M, Wright JJ, Allen SL, Kirschbaum MH, Zain J, Prince HM, Leonard JP, Geskin LJ, Reeder C, Joske D, Figg WD, Gardner ER, Steinberg SM, Jaffe ES, Stetler-Stevenson M, Lade S, Fojo AT, Bates SE. Phase II multi-institutional trial of the histone deacetylase inhibitor romidepsin as monotherapy for patients with cutaneous T-cell lymphoma. J Clin Oncol. 2009 Nov 10;27(32):5410-7. doi: 10.1200/JCO.2008.21.6150. Epub 2009 Oct 13. PMID 19826128
- [Result] Piekarz RL, Frye R, Prince HM, Kirschbaum MH, Zain J, Allen SL, Jaffe ES, Ling A, Turner M, Peer CJ, Figg WD, Steinberg SM, Smith S, Joske D, Lewis I, Hutchins L, Craig M, Fojo AT, Wright JJ, Bates SE. Phase 2 trial of romidepsin in patients with peripheral T-cell lymphoma. Blood. 2011 Jun 2;117(22):5827-34. doi: 10.1182/blood-2010-10-312603. Epub 2011 Feb 25. PMID 21355097
- [Derived] Shustov A, Coiffier B, Horwitz S, Sokol L, Pro B, Wolfson J, Balser B, Eisch R, Popplewell L, Prince HM, Allen SL, Piekarz R, Bates S. Romidepsin is effective and well tolerated in older patients with peripheral T-cell lymphoma: analysis of two phase II trials. Leuk Lymphoma. 2017 Oct;58(10):2335-2341. doi: 10.1080/10428194.2017.1295143. Epub 2017 Mar 7. PMID 28264616
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-C-0049.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 7 cohorts were written in the protocol, the cohorts were consolidated for submission to the Food and Drug Administration (FDA) into the peripheral T-cell lymphoma (PTCL) and cutaneous T-cell lymphoma (CTCL) groups, thus they are presented in this format.
Period: Overall Study
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
Started | 47 | 84
Completed | 45 | 73
Not Completed | 2 | 11
Not completed — Refused further treatment | 0 | 7
Not completed — Switched to alternative treatment | 0 | 3
Not completed — Intercurrent illness | 1 | 0
Not completed — Death on study | 1 | 1

BASELINE CHARACTERISTICS:
Population: Although 7 cohorts were written in the protocol, the cohorts were consolidated for submission to the Food and Drug Administration (FDA) into the peripheral T-cell lymphoma (PTCL) and cutaneous T-cell lymphoma (CTCL) groups, thus they are presented in this format.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Total
Number analyzed (Participants) | 47 | 84 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 57 | 88
  >=65 years | 16 | 27 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.97 (12.56) | 57.85 (13.08) | 58.25 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 25 | 57 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 46 | 80 | 126
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 17 | 21
  White | 40 | 65 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 39 | 55 | 94
  Australia | 8 | 29 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: A rigorous composite assessment was employed with uni-dimensional measurements of skin and visceral disease sites assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) required clearing of all known disease sites. Partial response (PR) required documented response in skin (≥ 30% per RECIST) or lymph nodes (≥ 50% per the International Working Group (IWG) criteria, with response in both compartments for a determination of PR, IWG guidelines. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Progressive disease (PD) is at least a 20% increase in the sum of the target lesions, or the appearance of one or more new lesions. Lymph node disease was assessed bi-dimensionally using the IWG criteria. Bone marrow involvement, as recommended by IWG criteria, and presence of circulating malignant T-cells ascertained by flow cytometry.
Time Frame: up to 56.5 days
Population: Two participants were excluded. After further analysis it was determined that the participants did not have PTCL but a different form of lymphoma that was not known at the onset of enrollment.
Measure: Number; unit: participants
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
Number analyzed (Participants) | 45 | 84
participants
  Complete Response + Partial Response | 17 | 28
  Complete Response | 8 | 5
  Partial Response | 9 | 23
  Stable Disease | 5 | 32
  Progressive disease | 18 | 18
  Not Evaluable | 5 | 6

2. Primary Outcome: Duration of Response (DOR)
Description: DOR is defined as the date response was noted until disease was no longer considered to be responding. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria and the International Working Group Criteria (IWG).Complete response (CR) required clearing of all known disease sites. Partial response (PR) required documented response in skin (≥ 30% per RECIST) or lymph nodes (≥ 50% per the International Working Group (IWG) criteria, with response in both compartments for a determination of PR, IWG guidelines. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Progressive disease (PD) is at least a 20% increase in the sum of the target lesions, or the appearance of one or more new lesions. Lymph node disease was assessed bi-dimensionally using the IWG criteria. Bone marrow involvement, as recommended by IWG criteria, and presence of circulating malignant T-cells ascertained by flow cytometry.
Time Frame: up to 127 months
Measure: Median (Full Range); unit: Months
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
Number analyzed (Participants) | 47 | 84
Months
  Complete Response/Partial Response | 9 [2 to 76] | 13.8 [1 to 127]
  Complete Response | 74 [3 to 76] | 19.3 [8 to 127]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 147 months and 5 days
Measure: Number; unit: participants
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
Number analyzed (Participants) | 47 | 84
participants | 47 | 84
Statistical Analysis 1: Comparison: Peripheral T-cell Lymphoma (PTCL) vs Cutaneous T-cell Lymphoma (CTCL); Test type: Superiority or Other; p < 0.01, Cochran-Armitage trend test — An exact Cochran-Armitage trend test was used to compare the distributions. In view of the large number of tests performed, we only refer to those with P-values <0.01 as statistically significant, with those for which 0.01 <P< 0.05 considered trends

4. Secondary Outcome: Median Number of Cycles of Depsipeptide Administered
Description: Participants were administered Depsipeptide and cycles (each cycle is 21 days) were monitored from the prescribed dose or higher to determine reductions (if needed) to maintain tolerability.
Time Frame: 83 cycles (i.e., each cycle is 21 days)
Measure: Median (Full Range); unit: Cycles per patient
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
Number analyzed (Participants) | 47 | 84
Cycles per patient | 3 [1 to 83] | 4.5 [1 to 79]

5. Secondary Outcome: Time to Progression
Description: Time to progression is defined from the first day of therapy until documentation of progressive disease. Progressive disease (PD) is at least a 20% increase in the sum of the target lesions, or the appearance of one or more new lesions. Lymph node disease was assessed bi-dimensionally using the International Working Group (IWG) criteria. Bone marrow involvement, as recommended by IWG criteria, and presence of circulating malignant T-cells ascertained by flow cytometry.
Time Frame: Until disease progression, or 30 days following off study date
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
Number analyzed (Participants) | 47 | 94
Months | 4.8 [2.0 to 9.3] | 6.4 [3.9 to 11.3]

6. Secondary Outcome: Fold Change in Histone Acetylation
Description: Fold change is calculated by dividing the level of histone acetylation in a treated sample (at 4, 24, and 48 hours) measured as intensity on a dot blot immunoassay, divided by the intensity in the pre-treatment sample. We considered a ≥ 2-fold change a measurable difference, and indicative of successful HDAC inhibition by romidepsin (depsipeptide).
Time Frame: 4 hours, 24 hours, and 48 hours after Romidepsin
Population: Global histone acetylation of all samples at pretreatment was designated as 1; values at other time points for each patient were calculated relative to the corresponding pretreatment value.
Measure: Median (Full Range); unit: Fold change
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
Number analyzed (Participants) | 18 | 29
Fold change
  4 hours | 2.99 [0.53 to 11.03] | 3.00 [0.44 to 17.30]
  24 hours | 1.97 [0.67 to 6.71] | 1.78 [0.037 to 17.45]
  48 hours | 0.62 [0.22 to 1.02] | 1.67 [0.28 to 17.64]

7. Secondary Outcome: Multidrug Resistance Protein 1 (MDR1) or ATP-binding Cassette Sub-family B Member 1 (ABCB1) Gene Expression
Description: Total ribonucleic acid (RNA) was isolated from peripheral blood mononuclear cells or patient tissue biopsies and analyzed by quantitative polymerase chain reaction (qPCR). Expression of MDR-1/ABCB1 was determined by qPCR relative to an RNA standard, then normalized to ribosomal RNA (rRNA). Fold change is calculated by dividing the level of MDR-1 in a treated sample (at 4, 24, and 48 hours) measured by qPCR, divided by MDR-1 in the pre-treatment sample. We considered a ≥ 2-fold change a measurable difference, and indicative of successful HDAC inhibition by romidepsin (depsipeptide).
Time Frame: 4 hours, 24 hours, and 48 hours after Romidepsin
Population: ABCB1 expression of all samples at pretreatment was designated as 1; values at other time points for each patient were calculated relative to the corresponding pretreatment value.
Measure: Median (Full Range); unit: Fold change
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
Number analyzed (Participants) | 17 | 35
Fold change
  4 hours | 2.74 [1.62 to 5.50] | 1.78 [0.19 to 21.08]
  24 hours | 1.5 [0.053 to 3.4] | 1.53 [0.15 to 7.55]
  48 hours | 0.545 [0.53 to 0.56] | 1.205 [0.15 to 19.42]

ADVERSE EVENTS:
Time Frame: 147 months and 5 days
Description: Although 7 cohorts were written in the protocol, the cohorts were consolidated for submission to the Food and Drug Administration (FDA) into the peripheral T-cell lymphoma (PTCL) and cutaneous T-cell lymphoma (CTCL) groups, thus they are presented in this format.
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL)
All-Cause Mortality (participants affected / at risk) | 6/47 | 5/84
Serious Adverse Events (participants affected / at risk) | 20/47 | 38/84
Other Adverse Events (participants affected / at risk) | 47/47 | 83/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral T-cell Lymphoma (PTCL) (N=47) | Cutaneous T-cell Lymphoma (CTCL) (N=84)
ANC (absolute neutrophil count) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Death/ARDS (acute respiratory distress syndrome) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Death/Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac troponin T (Cardiac disorders) | 0 (0) | 1 (1)
Catheter-related infection (Infections and infestations) | 0 (0) | 2 (2)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
DOE (dyspnea on exertion) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Infection: EBV (Epstein Barr virus) reactivation (Infections and infestations) | 0 (0) | 1 (1)
Death/Infection with unknown ANC (absolute neutrophil count) (Infections and infestations) | 0 (0) | 1 (1)
Death/Infection without neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 4 (4) | 21 (25)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 0 (0) | 3 (3)
Death/Fever/Neutropenia (General disorders) | 0 (0) | 1 (1)
Fever/neutropenia (General disorders) | 0 (0) | 1 (1)
Fever without neutropenia (General disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgery:GI (gastrointestinal) intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
SVT (supraventricular tachycardia) (Cardiac disorders) | 1 (1) | 2 (2)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Wound infectious (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Infection: septic arthritis (Infections and infestations) | 0 (0) | 1 (1)
Bili increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death related to 2nd cancer:EBV (Epstein Barr virus) lymphoma (General disorders) | 1 (1) | 0 (0)
Death:cardiac arrest (General disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 4 (4) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection with grade 3 or 4 ANC (Infections and infestations) | 2 (2) | 0 (0)
Infection:catheter (Infections and infestations) | 1 (1) | 0 (0)
Melana (Gastrointestinal disorders) | 1 (1) | 0 (0)
Platelet (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Prolonged QTc (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Death progressive disease (General disorders) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral T-cell Lymphoma (PTCL) (N=47) | Cutaneous T-cell Lymphoma (CTCL) (N=84)
Anemia (Blood and lymphatic system disorders) | 38 (151) | 53 (166)
Anorexia (Gastrointestinal disorders) | 31 (124) | 37 (79)
Constipation (Gastrointestinal disorders) | 17 (29) | 33 (61)
Fatigue (General disorders) | 34 (129) | 68 (194)
Headache (Nervous system disorders) | 17 (32) | 18 (33)
Hyperglycemia (Metabolism and nutrition disorders) | 28 (127) | 33 (109)
Hypokalemia (Metabolism and nutrition disorders) | 14 (19) | 14 (35)
Hypermagnesemia (Metabolism and nutrition disorders) | 11 (67) | 21 (71)
Hyperuricemia (Metabolism and nutrition disorders) | 16 (86) | 25 (71)
Hyponatremia (Metabolism and nutrition disorders) | 15 (27) | 14 (26)
Hypotension (Cardiac disorders) | 12 (39) | 19 (42)
Lymphocyte count (Blood and lymphatic system disorders) | 0 (0) | 42 (149)
Nausea (Gastrointestinal disorders) | 38 (224) | 67 (266)
Neutrophil count (Blood and lymphatic system disorders) | 0 (0) | 44 (172)
Hypoalbuminemia (Hepatobiliary disorders) | 32 (146) | 36 (89)
Hypocalcemia (Metabolism and nutrition disorders) | 34 (142) | 37 (134)
Dysgeusia (Gastrointestinal disorders) | 20 (86) | 27 (54)
Hypophosphatemia (Metabolism and nutrition disorders) | 17 (55) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 36 (244) | 48 (300)
Diarrhea (Gastrointestinal disorders) | 17 (82) | 24 (44)
Fever (General disorders) | 18 (50) | 20 (45)
Vomiting (Gastrointestinal disorders) | 23 (101) | 40 (101)
Bilirubin increased (Hepatobiliary disorders) | 11 (76) | 18 (44)
Hypomagnesemia (Metabolism and nutrition disorders) | 16 (52) | 24 (68)
AST (aspartate transaminase)/SGOT (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 17 (58) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 7 (14)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Activated PTT (partial thromboplastin time) (Blood and lymphatic system disorders) | 0 (0) | 5 (7)
Acute kidney injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALT (alanine aminotransferase) (Hepatobiliary disorders) | 0 (0) | 22 (45)
Alk phos (Hepatobiliary disorders) | 0 (0) | 11 (23)
Allergic reaction (Immune system disorders) | 1 (1) | 4 (6)
Allergic rhinitis (Immune system disorders) | 4 (22) | 6 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 7 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
AST (aspartate aminotransferase) (Hepatobiliary disorders) | 0 (0) | 26 (68)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac disorder:T wave (Cardiac disorders) | 40 (514) | 57 (424)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Catheter-related infection (Infections and infestations) | 2 (2) | 5 (5)
Chills (General disorders) | 4 (4) | 6 (10)
Phlebitis (Cardiac disorders) | 0 (0) | 4 (4)
Cholesterol high (Metabolism and nutrition disorders) | 1 (1) | 4 (8)
Conduction disorder (Cardiac disorders) | 0 (0) | 3 (3)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 7 (17)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 5 (6) | 11 (20)
Creatinine increased (Renal and urinary disorders) | 10 (26) | 11 (14)
Dehydration (Gastrointestinal disorders) | 4 (8) | 8 (11)
Depression (Nervous system disorders) | 4 (4) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5) | 8 (15)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Dyspepsia on exertion (Gastrointestinal disorders) | 0 (0) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 13 (19)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 5 (8)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Eye disorder (Eye disorders) | 0 (0) | 6 (6)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Infections and infestations) | 0 (0) | 2 (3)
Flushing (Skin and subcutaneous tissue disorders) | 2 (7) | 3 (3)
GERD (gastroesophageal reflux disease) (Gastrointestinal disorders) | 0 (0) | 4 (4)
GGT (gamma glutamyltransferase) increased (Hepatobiliary disorders) | 0 (0) | 4 (9)
Hematuria (Renal and urinary disorders) | 2 (3) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Viral hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hot flashes (Endocrine disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (18) | 5 (37)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (15) | 8 (13)
Hypernatremia (Metabolism and nutrition disorders) | 3 (7) | 3 (7)
Hypertension (Cardiac disorders) | 1 (3) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 8 (11) | 9 (23)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 16 (45)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infections (Infections and infestations) | 18 (38) | 22 (75)
INR (International Normalized Ratio) increased (Investigations) | 2 (2) | 4 (11)
Insomnia (Nervous system disorders) | 4 (4) | 5 (7)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Lower GI hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 6 (9)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 5 (8)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Non cardiac chest pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (6)
Oral pain/mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 10 (24) | 21 (25)
Palpitations (Cardiac disorders) | 1 (2) | 4 (4)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 7 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 12 (14) | 22 (35)
Psychosis (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash-maculo-papular (Skin and subcutaneous tissue disorders) | 12 (15) | 23 (26)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
UTI (urinary tract infection) (Renal and urinary disorders) | 0 (0) | 6 (14)
Vaginal mucositis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
URI (upper respiratory infection) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Sinus bradycardia (Cardiac disorders) | 4 (4) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SVT (supraventricular tachycardia) (Cardiac disorders) | 2 (3) | 3 (5)
Syncope (Nervous system disorders) | 1 (1) | 3 (5)
Thromboembolic event (Vascular disorders) | 1 (1) | 4 (4)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 7 (9)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 4 (5)
Ventricular arrhythmia (Cardiac disorders) | 3 (5) | 2 (3)
Vision changes (Eye disorders) | 0 (0) | 1 (1)
Voice alteration/hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Weight gain (General disorders) | 0 (0) | 1 (1)
Weight loss (General disorders) | 6 (6) | 11 (15)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
WBC (white blood cell) decreased (Blood and lymphatic system disorders) | 31 (195) | 35 (136)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urine incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Serum amylase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lipase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (7) | 0 (0)
Euphoria (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 3 (4) | 0 (0)
Alkalosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 2 (9) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Troponin I increased (Cardiac disorders) | 1 (1) | 0 (0)
Troponin T increased (Cardiac disorders) | 1 (1) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 5 (8) | 4 (4)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 26 (105) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 35 (211) | 0 (0)
ALT(alanine aminotransferase)/SGPT (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 15 (53) | 0 (0)
Alkaline phosphokinase increased (Hepatobiliary disorders) | 5 (8) | 0 (0)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
7 cohorts were consolidated for submission to the Food and Drug Administration (FDA) into the peripheral T-cell lymphoma (PTCL) and cutaneous T-cell lymphoma (CTCL) groups, thus they are presented in this format.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No